CLINICAL TRIAL: NCT00746252
Title: Investigating Metabolic Side Effects of Antipsychotic Medications in Children
Brief Title: Side Effect Study of Antipsychotic Medicines to Treat Childhood Bipolar Disorder
Acronym: PAMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due low rate of participation and lack of funding
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Gloria Reeves, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00043695
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2018-03-21 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Bipolar Disorder
Keywords: bipolar; children; antipsychotic; side effect
MeSH Terms: conditions — Bipolar Disorder | interventions — Risperidone; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): risperidone
  Interventions: Drug: risperidone
- 2 (Experimental): aripiprazole
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: risperidone — Children will have a flexible dose titration based on their unique response to the medication (assessed using clinical global improvement scores). Children will be treated for six months using daily, bid dosing.
  Other Names: Brand name: Risperdal
  Arms: 1
Drug: aripiprazole — children will have a flexible dosing titration based on their unique response (assessed using clinical global improvement scores). Children will be treated with daily medication for six months.
  Other Names: Brand name: Abilify
  Arms: 2

SUMMARY:
The purpose of this study is to learn more about weight gain and related side effects when children are treated with antipsychotic medicine for mood disorders.

DETAILED DESCRIPTION:
This protocol is a six month, randomized, open label trial of risperidone versus aripiprazole in antipsychotic naive youth (7 - 12 years old) who have been identified by their clinical treatment provider as needing antipsychotic treatment of a bipolar disorder.

This study proposes to monitor changes in metabolic parameters (body mass index percentile, % body fat, insulin resistance, and lipid levels) over the course of six months treatment with aripiprazole or risperidone in youth with a bipolar spectrum disorder. We will also assess possible mechanisms of second generation antipsychotic induced weight gain by monitoring physical activity and hunger/appetite changes over the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* We will include children, ages 7 - 12 years old, male and female with diagnosis of a bipolar spectrum disorder.
* Specific diagnoses included are as follows:

  * Bipolar I disorder,
  * Bipolar II disorder,
  * Bipolar Disorder Not Otherwise Specified,
  * Mood Disorder Not otherwise specified.
* The inclusion of a spectrum of bipolar diagnosis is because children with moderate to severe impairment from mood symptoms often still do not meet criteria for Bipolar I disorder since young children tend to have more chronic (non-episodic) course of symptoms and diagnostic criteria for Bipolar I disorder are more difficult to apply to adults than young children (e.g. symptoms of grandiosity and euphoria).
* No prior treatment with an antipsychotic medication for >30 days. This criteria was added because weight loss on an assigned treatment may be due to discontinuing a prior antipsychotic medication rather than due to the current treatment.
* Recommendation from a current psychiatric treatment provider for treatment with an antipsychotic medication.
* This inclusion criteria provides an added layer of safety in that youth who have referred for the study have already been deemed by their independent provider to need an antipsychotic medication, so we are only exposing children to antipsychotic treatment who would have been treated with this type of medication regardless of whether or not there care was provided in a research or clinical program.

Exclusion Criteria:

* Medications: We will exclude children who are on current treatment with

  * oral steroids,
  * lithium,
  * depakote since these medications will have a confounding effect on weight.
* We will allow children on stimulant medication to participate, because ADHD comorbidity is very high in prepubertal bipolar disorder (unlike adolescent or adult onset bipolar disorder).
* We are including ADHD children to thus increase generalizability of the study, and it would be inappropriate to withhold stimulant treatment from these children for a six month period.
* Recruitment will be stratified to make sure there are equal numbers of patients on stimulants in each group.
* Somatic Conditions: We will exclude children with diabetes (type I or type II), and those with physical disability that would interfere with physical activity (will specifically exclude children whose guardian reports that the child has been medically excused from physical education at their school program because of physical disability) since insulin sensitivity and activity levels are outcome measures being assessed in this protocol.
* We will exclude youth with mental retardation, by parent report. Cognitive screening will be done with the Wechsler Abbreviated Scale of Intelligence (WASI).
* Youth with an IQ less than 70 will be excluded because they may have difficulty with self report measures.
* We will exclude children who have a history of treatment of an antipsychotic medication for >30 days, as explained above.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Reeves, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, School of Medicine, Department of Psychiatry, Division of Child and Adolescent Psychiatry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants enrolled and completed baseline assessments but were withdrawn from the study at baseline due to the following reasons:
  1. Abnormal glucose tolerance test requiring further assessment with endocrinology.
  2. Unable to complete lab work due to increased distress.
Groups:
- Risperidone: risperidone
  risperidone: Children will have a flexible dose titration based on their unique response to the medication (assessed using clinical global improvement scores). Children will be treated for six months using daily, bid dosing.
- Aripiprazole: aripiprazole
  aripiprazole: children will have a flexible dosing titration based on their unique response (assessed using clinical global improvement scores). Children will be treated with daily medication for six months.
Period: Overall Study
Arm/Group | Risperidone | Aripiprazole
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — weight gain >7.5 % | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone | Aripiprazole | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.75 (0) | 12.5 (0) | 10.9 (2.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain
Description: Weight gain from baseline to last observation up to 12 weeks. Last observation carried to 12 weeks.
Time Frame: These measurements are done biweekly from baseline up until 12 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Risperidone | Aripiprazole
Number analyzed (Participants) | 1 | 2
pounds | 8.5 (NA) — Unable to calculate SD for 1 participant. | 6.65 (1.48)
Statistical Analysis 1: Comparison: Risperidone vs Aripiprazole; Comparison of mean weight gain between groups; Test type: Other; p = .495, t-test, 2 sided — Threshold of significance is p<.05

ADVERSE EVENTS:
Arm/Group | Risperidone | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone (N=1) | Aripiprazole (N=2)
Weight gain (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — The protocol stopping criteria was if the participant had an increase in weight that exceeded 5% of their baseline weight.

LIMITATIONS AND CAVEATS:
The study funding stopped before a sufficient number of participants could be enrolled and therefore the study was terminated. Additionally the stopping criteria of 5% weight gain limited the length of time participants were in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No